CLINICAL TRIAL: NCT07228416
Title: Milky Way Sensor: Device Validation for Non-Infiltrated Tissues
Brief Title: Milky Way Sensor Motion Validation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVW-CLR-CS37-400
Record Dates: First submitted 2025-11-12; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Infiltration of Peripheral IV Therapy
Keywords: motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Non-Infiltrated Tissue (Experimental): The ivWatch Model 400 monitored a common peripheral IV site over a 24 hour observation period.
  Interventions: Device: ivWatch Model 400

INTERVENTIONS:
Device: ivWatch Model 400 — The ivWatch Model 400 monitored tissue at common IV sites over a 24 hour period.

SUMMARY:
A single arm study of 20 adult volunteers to assess the safety and efficacy of the ivWatch sensors when observing non-infiltrated (normal) tissues at common peripheral IV therapy sites.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Healthy individual, verified by an eligible designation on the Health History Form

Exclusion Criteria:

* Currently enrolled in another clinical trial
* Currently pregnant or trying to become pregnant
* Serious and uncontrolled medical condition
* Tattoo(s), scarring, or bruising that severely limits vein visualization at a sensor monitoring location
* Medical adhesive allergy
* Sleepwalking occurrence in the last year
* Current drug/alcohol dependence
* Sick or had an infection in the last 14 days
* Hospitalized in the last 14 days
* Fever at the time of study visit (≥100.4°F)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Check IV notification rate per day | 24 Hours
  The ivWatch Model 400 issues Check IV notifications to communicate the need for a clinician to check an IV site. A red notification suggests an increased likelihood that an IV infiltration may be occurring, with a greater likelihood relative to a yellow notification. This measure describes the average number of red notifications issued by the ivWatch device in a given day when monitoring normal, non-infiltrated tissues. The 95% confidence interval for the red notification rate was calculated using a negative binomial regression model.